CLINICAL TRIAL: NCT05589454
Title: Intracranial Hemorrhage Risk of Intensive Statin Therapy in Patients With Acute Ischemic Stroke Combined With Cerebral Microbleeds
Brief Title: Intracranial Hemorrhage Risk of Intensive Statin in Acute Ischemic Stroke With Cerebral Microbleeds
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sichuan Provincial People's Hospital (Other)
Collaborators: Science and Technology Department of Sichuan Province (Other)
Responsible Party: Principal Investigator, Jialing Zhao, Principal Investigator, Sichuan Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: zjl8803302022NSCSC1374
Record Dates: First submitted 2022-10-11; First posted 2022-10-21 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Acute Ischemic Stroke; Cerebral Microbleeds
Keywords: Acute Ischemic Stroke; Intracranial Hemorrhage Risk; Cerebral Microbleeds; Intensive Statin Therapy
MeSH Terms: conditions — Ischemic Stroke | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-dose atorvastatin (Experimental): atorvastatin calcium tablets 80 mg, quaque nocte, continue to the end of the study
  Interventions: Drug: Atorvastatin Calcium tablets 80mg
- Low-dose atorvastatin (Active Comparator): atorvastatin calcium tablets 20 mg, quaque nocte, continue to the end of the study
  Interventions: Drug: Atorvastatin Calcium tablets 20mg

INTERVENTIONS:
Drug: Atorvastatin Calcium tablets 80mg — Atorvastatin calcium tablets 4 pills (80 mg) will be given at a fixed time every night (24 ± 1 h between two doses) , orally, until the end of follow-up
  Other Names: ALe produced by Jialin pharmaceutical company
  Arms: High-dose atorvastatin
Drug: Atorvastatin Calcium tablets 20mg — Atorvastatin calcium tablets 1 pill (20 mg) will be given at a fixed time every night (24 ± 1 h between two doses) , orally, until the end of follow-up
  Other Names: ALe produced by Jialin pharmaceutical company
  Arms: Low-dose atorvastatin

SUMMARY:
This study is the first and largest secondary prevention trial about lipid-lowering therapy for acute ischemic stroke patients at high-risk of intracranial hemorrhage.

The primary hypothesis of this study is: excessive reduction in serum lipid levels by intensive statin therapy in acute ischemic stroke patients with cerebral microbleeds can increase the risk of intracranial hemorrhage.

This study will shed light on new clinical decisions regarding the long-term serum lipid management in these patients with dilemma in clinical practice.

DETAILED DESCRIPTION:
Cerebral microbleeds are an important subtype of cerebral small vessel diseases that have been established in approximately one third of patients with ischemic stroke and are associated with the risk of recurrent ischemic stroke, symptomatic intracranial hemorrhage, and all-cause death. In patients with ischemic stroke or transient ischemic attack, the relative and absolute risks of intracranial hemorrhage increase more rapidly than the risk of ischemic stroke with the increase of cerebral microbleeds burden, but the absolute incidence of ischemic stroke is still higher than that of cerebral hemorrhage.

It has been generally accepted that statins can effectively prevent recurrent ischemic stroke by reducing serum lipid levels. However, both low serum lipid levels and high dose of statins are clear risk factors for intracerebral hemorrhage, and the reduction of major serum lipid levels may increase the risk of cerebral microbleeds. Of note, the risk of statin mediated hemorrhage appears to depend on the degree of lipid reduction rather than statin use per se. These observations raise concerns about the safety of lipid-lowering therapy, especially intensive lipid-lowering therapy, in patients with acute ischemic stroke and cerebral microbleeds who are at high risk for future intracranial hemorrhage. It is still not clear that how to carry on the proper management of serum lipid levels in this particular population to reduce the recurrence of ischemic events as well as hemorrhagic events, for there is still a lack of clinical studies to explore the risk and benefit of different doses of statins to achieve different degrees of lipid regulation.

So, if it is proved that excessive reduction in serum lipid levels by intensive statin therapy in acute ischemic stroke patients with cerebral microbleeds can increase the risk of future intracranial hemorrhage, we will inform new clinical decisions regarding the long-term lipid management in these patients with dilemma in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a non-cardioembolic ischemic stroke within 14 days prior to entry to the study
2. Adults between the ages of 18 and 85
3. Patients with cerebral microbleeds on baseline SWI imaging
4. Patients or their legal representatives volunteer to participate and sign written informed consent

Exclusion Criteria:

1. Patients with severe acute ischemic stroke (NIHSS score ≥21)
2. Patients with coma (GCS score < 8)
3. Patients with previous moderate to severe dependence (mRS score 3-5)
4. Patients with any contraindications to CT and MRI (such as metal implants, claustrophobia, etc.)
5. Patients who are allergic to atorvastatin or excipients
6. Patients with intracranial hemorrhagic diseases confirmed by CT or MRI, such as cerebral hemorrhage, epidural hematoma, subdural hematoma, ventricular hemorrhage, subarachnoid hemorrhage, traumatic cerebral hemorrhage or hemorrhagic conversion of infarcts, etc
7. Patients within 6 months after hemorrhagic stroke
8. Patients with hemorrhagic tendency, such as abnormal coagulation function, Henoch-Schonlein purpura, platelet count less than 100×109/L or abnormal platelet function, etc
9. Patients who are ready to undergo or have undergone intravenous thrombolysis after the onset of the disease or who require urgent or recent (within 90 days) endovascular treatment;
10. Patients with severe hypertension (systolic blood pressure ≥ 185 mmHg or diastolic blood pressure ≥ 110 mmHg) that has not been controlled by treatment
11. Patients with hypoglycemia (< 2.7 mmol/L) or hyperglycemia (>22.2 mmol/L)
12. Patients with previous cerebral arteritis, brain tumor, cerebral parasitic disease, cerebral arteriovenous malformation, cerebral cavernous hemangioma, cerebral aneurysm, severe craniocerebral injury, or intracranial infection
13. Patients with previous severe valvular heart disease, atrial fibrillation, acute myocardial infarction or interventional therapy in the past 6 months, heart failure (patients classified as class III-IV according to the New York Heart Association [NYHA]) or patients with indications for pacemaker placement but without pacemaker installation or other malignant arrhythmias
14. Patients contraindicate to antiplatelet therapy;
15. Patients who must use other types of statins or other types of lipid-lowering drugs such as ezetimibe
16. Patients with severe mental disorders or dementia that are unable or unwilling to cooperate
17. Patients with active liver disease or unexplained 2 or more abnormal liver function tests (alanine aminotransferase [ALT] or aspartate aminotransferase [AST] ≥ 3.0× upper limit of normal [ULN])
18. Patients with myositis, myopathy, rhabdomyolysis, or 2 or more episodes of unexplained serum creatine kinase[CK] elevation ([CK]≥5.0×ULN)
19. Patients with other serious systemic or organic diseases that investigators believe will not allow evaluation of efficacy or are unlikely to complete the expected course of treatment and follow-up (e.g., malignancy, life expectancy < 3 years, etc.)
20. Women who are pregnant, breastfeeding or planning to become pregnant and who do not want to use contraception
21. Patients who participated in or are participating in other clinical trials during the 3 months prior to the study
22. Patients who are deemed ineligible for clinical trial participation by the investigator
23. Patients or their legal representatives do not consent to participate in this study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
The incidence of hemorrhagic strokes | From date of randomization until the date of the first occurrence of hemorrhagic stroke, assessed up to 36 months
Changes in degree of cerebral microbleeds | From date of randomization until the end of the study, assessed up to 36 months
  The degree is divided into: mild (1-2), moderate (3-10), severe (more than 10), calculate and compare the proportions of different degrees at baseline and the end of the study

SECONDARY OUTCOMES:
The Incidence of recurrent ischemic stroke and transient ischemic attack | From date of randomization until the date of the first recurrent of ischemic stroke or the first occurrence of transient ischemic attack, assessed up to 36 months
The Incidence of myocardial infarction | From date of randomization until the date of the first occurrence of myocardial infarction, assessed up to 36 months
The Incidence of cardiovascular death | From date of randomization until the date of cardiovascular death, assessed up to 36 months
The mean of serum triglycerides (TG) levels | From date of randomization until the end of the study, assessed up to 36 months
  Calculate the mean of serum TG levels for 3 years with at least 3 measurements
The mean of serum total cholesterol (TC) levels | From date of randomization until the end of the study, assessed up to 36 months
  Calculate the mean of serum TC levels for 3 years with at least 3 measurements
The mean of serum low-density lipoprotein cholesterol (LDL-C) levels | From date of randomization until the end of the study, assessed up to 36 months
  Calculate the mean of serum LDL-C levels for 3 years with at least 3 measurements
The mean of serum high-density lipoprotein cholesterol (HDL-C) levels | From date of randomization until the end of the study, assessed up to 36 months
  Calculate the mean of serum HDL-C levels for 3 years with at least 3 measurements
The variability of serum triglycerides (TG) levels | From date of randomization until the end of the study, assessed up to 36 months
  Calculate the variability of serum TG levels for 3 years with at least 3 measurements
The variability of serum total cholesterol (TC) levels | From date of randomization until the end of the study, assessed up to 36 months
  Calculate the variability of serum TC levels for 3 years with at least 3 measurements
The variability of serum low-density lipoprotein cholesterol (LDL-C) levels | From date of randomization until the end of the study, assessed up to 36 months
  Calculate the variability of serum LDL-C levels for 3 years with at least 3 measurements
The variability of serum high-density lipoprotein cholesterol (HDL-C) levels | From date of randomization until the end of the study, assessed up to 36 months
  Calculate the variability of serum HDL-C levels for 3 years with at least 3 measurements
The proportions of different degrees of CMBs at the end of the study | From date of randomization until the end of the study, assessed up to 36 months
  Calculate the proportions of different degrees of CMBs (mild, moderate and severe) at the end of the study
The correlation between the mean of serum triglycerides (TG) levels and the proportions of different degrees of CMBs | From date of randomization until the end of the study, assessed up to 36 months
The correlation between the mean of serum total cholesterol (TC) levels and the proportions of different degrees of CMBs | From date of randomization until the end of the study, assessed up to 36 months
The correlation between the mean of serum low-density lipoprotein cholesterol (LDL-C) levels and the proportions of different degrees of CMBs | From date of randomization until the end of the study, assessed up to 36 months
The correlation between the mean of serum high-density lipoprotein cholesterol (HDL-C) levels and the proportions of different degrees of CMBs | From date of randomization until the end of the study, assessed up to 36 months
The correlation between the variability of serum triglycerides (TG) levels and the proportions of different degrees of CMBs | From date of randomization until the end of the study, assessed up to 36 months
The correlation between the variability of serum total cholesterol (TC) levels and the proportions of different degrees of CMBs | From date of randomization until the end of the study, assessed up to 36 months
The correlation between the variability of serum low-density lipoprotein cholesterol (LDL-C) levels and the proportions of different degrees of CMBs | From date of randomization until the end of the study, assessed up to 36 months
The correlation between the variability of serum high-density lipoprotein cholesterol (HDL-C) levels and the proportions of different degrees of CMBs | From date of randomization until the end of the study, assessed up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Jialing Zhao, MD, Principal Investigator — Departement of Neurology, Sichuan Academy of Medical Sciences & Sichuan Provincial People's Hospital; Yang Xiang, MD, Study Director — Departement of Neurology, Sichuan Academy of Medical Sciences & Sichuan Provincial People's Hospital
Locations (5):
- China (5):
  - Yunyang County People's Hospital, Chongqing, Chongqing Municipality
  - Chengdu Eighth People's Hospital, Chengdu, Sichuan
  - Sichuan Academy of Medical Sciences & Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Ya 'an People's Hospital, Ya'an, Sichuan
  - Zigong Third People's Hospital, Zigong, Sichuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhao JL, Ai CB, Wang L, Yang SJ, Wang J, Yang W, Tang J, Zhang L, Li Y, Yan TQ, Gou S, Xie GG, Xiang Y. A multicenter, prospective, randomized controlled trial of intracranial hemorrhage risk of intensive statin therapy in patients with acute ischemic stroke combined with cerebral microbleeds (CHRISTMAS): Study protocol. Front Neurol. 2023 Feb 9;14:1097078. doi: 10.3389/fneur.2023.1097078. eCollection 2023. PMID 36846138